CLINICAL TRIAL: NCT04665869
Title: Long-term Effects of Combined Balance and Brisk Walking on Alleviating Motor and Non-motor Symptoms in Parkinson's Disease: a Randomized Controlled Trial
Brief Title: Long-term Effects of Combined Balance and Brisk Walking in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Margaret Kit Yi Mak, Professor, Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20191206002
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: rehabilitation; aerobic exercise; postural balance
MeSH Terms: conditions — Parkinson Disease | interventions — Pliability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined balance and brisk walking training (Experimental): Week1-6: Supervised training in groups of 6-8 participant, once/week, 90 min/session 2. Week 7-26: Supervised training in groups of 6-8 participant, once/month, 90 min/session 3. Participants practice own balance exercise and brisk walking 2-3 times/week (to aim at 150 min of moderate intensity of brisk walking per week at 40-60% of heart rate reserve)
  Interventions: Behavioral: Combined balance and brisk walking training
- Flexibility and strengthening exercise (Active Comparator): 1. Week1-6: Supervised training in groups of 6-8 participant, once/week, 90 min/session
  2. Week 7-26: Supervised training in groups of 6-8 participant, once/month, 90 min/session
  3. Participants practice own flexibility and strengthening exercise 2-3 times/week (to aim at 150 min of exercise per week)
  Interventions: Behavioral: Flexibility and strengthening exercise

INTERVENTIONS:
Behavioral: Combined balance and brisk walking training — 6-months of combined balance and brisk walking training
  Arms: Combined balance and brisk walking training
Behavioral: Flexibility and strengthening exercise — 6-months of flexibility and strengthening exercise
  Arms: Flexibility and strengthening exercise

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disease characterized with both clinical motor and non-motor features, as well as decrease in balance performance and walking endurance. The non-motor symptoms such as depression, anxiety, sleep disturbance and fatigue wound impose negative impacts on the quality of life of the individuals with PD. Aerobic endurance training can improve physical capacity and reduce those non-motor symptoms such as mood and sleep disorders. Based on the results of our recent pilot study, brisk walking is a safe and moderate-level aerobic walking exercise for improving walking capacity in the PD population up to 6 week after treatment ended. Community-based balance training could also enhance balance performance and dual-task gait performance up to 12-month follow-up for people with PD. The primary purpose of this proposed study is to investigate the short- and long-term effects of a 6-month balance and brisk walking programme in alleviating non-motor and motor symptoms in people with PD. The secondary objective is to examine the short- and long-term effects of a 6-month balance and brisk walking program on enhancing walking capacity, balance performance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease diagnosed by neurologist with Hoehn & Yahr stage 2 or 3
* Having a 30-meter walking ability

Exclusion Criteria:

* Significant neurological condition (other than Parkinson's disease)
* Musculoskeletal conditions affecting gait, balance or functions
* Had received deep brain stimulation surgery
* Cognitive impairment with Montreal Cognitive Assessment score <24
* Present with on-off motor fluctuations.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society Unified Parkinson Disease Rating Scale Part III (MDS-UPDRS-III) score | 1 year
  This score consists of 18 items in 33 questions examining the motor and functional capacity of people with Parkinson's disease by the assessor. Each question will be rated from 0 (normal) to 4 (severe). The MDS-UPDRS-III score ranges from 0 to 132, with higher scores indicating more severe motor and functional impairments
Movement Disorder Society Unified Parkinson Disease Rating Scale Part I (MDS-UPDRS-I) score | 1 year
  This score assesses the non-motor aspects of experiences of daily living in people with Parkinson's disease with a total of 13 questions. The score will be administered by assessor asking participants about their behaviors and non-motor symptoms such as cognitive impairment, hallucination, depressive and anxious mood, sleep, pain, urinary and constipation problems, and fatigue etc. Each question will be rated from 0 (normal) to 4 (severe). The MDS-UPDRS-I score ranges from 0 to 52, with higher scores indicating more severe non-motor impairment.

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test (mini-Best) total score | 1-year
  To evaluate dynamic balance in four domains: anticipatory postural adjustments, postural reactions, sensory integration and gait stability. The mini-BEST total score ranges from 0 to 28, with a higher score indicates better dynamic balance.
Six-minute walking test (6MWT) distance | 1 year
  The maximum walking distance covered during a validated six-minute walk test (6MWT) to document participants' aerobic endurance level and walking capacity
Single-task timed-up-and-go (TUG) time | 1 year
  The single-task gait performance measured by the time taken to complete 3-meter timed-up-and-go (TUG) test
Dual-task timed-up-and-go (DTUG) time | 1 year
  The dual-task gait performance measured by the time taken to complete 3-meter timed-up-and-go test with serial subtraction
Five-times-sit-to-stand (FTSTS) time | 1 year
  The composite lower limb strength measured by the time taken to complete 5 repetitions of sitting to standing
Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) total score | 1 year
  The Non-Motor Symptoms Scale is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The NMSS total score ranges form 0 to 360, with a higher score indicates worse PD non-motor symptoms.
Gait cycle measures by 2-minute Instrument Walk Test using mobile sensors in both comfortable and fast walking speed | 1 year
  Spatial, gait phase, spatiotemporal and asymmetric walking variables such as gait speed, cadence, stride length, arm swing angle and velocity, and trunk movement angle and velocity will be measured by Mobility Lab system.
Activities-specific Balance Confidence (ABC) Scale score | 1 year
  The ABC score will be used to measure the participants' perceived level of balance confidence in 16 indoor and outdoor activities. Each activity is rated from 0-100 (0 indicates no confidence and 100 indicates full confidence, total score=1600). The total score is converted into percentage score ranging from 0 to 100%, with a higher ABC score indicating a higher level of balance confidence.
Parkinson Disease Questionnaire-39 (PDQ-39) summary index score | 1 year
  It is a health-related quality-of-life outcome measure that contains 39 self-reported items on eight domains, i.e.: mobility [#1-10], activities of daily living [#11-16], emotional well-being [#17-22], stigma [#23-26], social support [#27-29], cognition [#30-33], communication [#34-36], and body discomfort [#37-39]. The PDQ-39 has been translated into Chinese and validated for local use. Each item is scored on 5-point Likert-type scales ranging from 0 (never), 1 (occasionally), 2 (sometimes), and 3 (often) to 4 (always) based on their perception on the item over the past month. The PDQ-39 total score is 156 and the PDQ-39 summary index is created by summing all eight of the PDQ-39 domains and standardizing the score on a scale of 0-100%. A lower PDQ-39 summary index score reflects a better health-related quality-of-life.
Pittsburgh Sleep Quality Index (PSQI) | 1 year
  The Pittsburgh Sleep Quality Index is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score of "5" or greater is indicative of poor sleep quality.
Fall risk | 1 year
  The risk of falling of each group will be determined by the ratio of non-fallers to fallers at treatment completion and 6-month follow-up. A lower risk ratio indicates a lower risk of falling.
Fall rate | 1 year
  The fall rate (times of fall per year per person) of each group at treatment completion and 6-month follow-up will be calculated with the following formula:
  Number of fall events X12 / (Number of months spent to assemble fall data X number of subjects)
  A lower fall rate indicates a better effect on fall reduction.
Injurious fall risk | 1 year
  The risk of injurious falling of each group at treatment completion and 6-month follow-up will be determined by the ratio of injurious non-fallers to injurious fallers. A lower injurious risk ratio indicates a lower risk of injurious falling.
Injurious fall rate | 1 year
  The injurious fall rate (times of injurious fall per year per person) of each group at treatment completion and 6-month follow-up will be calculated with the following formula:
  Number of injurious fall events X12 / (Number of months spent to collect injurious fall data X number of subjects)
  A lower injurious fall rate indicates a better effect on injurious fall reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Mak, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Nothing Selected, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tysnes OB, Storstein A. Epidemiology of Parkinson's disease. J Neural Transm (Vienna). 2017 Aug;124(8):901-905. doi: 10.1007/s00702-017-1686-y. Epub 2017 Feb 1. PMID 28150045
- [Background] Mak MK, Wong-Yu IS, Shen X, Chung CL. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol. 2017 Nov;13(11):689-703. doi: 10.1038/nrneurol.2017.128. Epub 2017 Oct 13. PMID 29027544
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Benka Wallen M, Franzen E, Nero H, Hagstromer M. Levels and Patterns of Physical Activity and Sedentary Behavior in Elderly People With Mild to Moderate Parkinson Disease. Phys Ther. 2015 Aug;95(8):1135-41. doi: 10.2522/ptj.20140374. Epub 2015 Feb 5. PMID 25655884
- [Background] Seppi K, Weintraub D, Coelho M, Perez-Lloret S, Fox SH, Katzenschlager R, Hametner EM, Poewe W, Rascol O, Goetz CG, Sampaio C. The Movement Disorder Society Evidence-Based Medicine Review Update: Treatments for the non-motor symptoms of Parkinson's disease. Mov Disord. 2011 Oct;26 Suppl 3(0 3):S42-80. doi: 10.1002/mds.23884. PMID 22021174
- [Background] Reynolds GO, Otto MW, Ellis TD, Cronin-Golomb A. The Therapeutic Potential of Exercise to Improve Mood, Cognition, and Sleep in Parkinson's Disease. Mov Disord. 2016 Jan;31(1):23-38. doi: 10.1002/mds.26484. Epub 2015 Dec 30. PMID 26715466
- [Background] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037
- [Background] Tully MA, Cupples ME, Chan WS, McGlade K, Young IS. Brisk walking, fitness, and cardiovascular risk: a randomized controlled trial in primary care. Prev Med. 2005 Aug;41(2):622-8. doi: 10.1016/j.ypmed.2004.11.030. PMID 15917061
- [Background] Wong-Yu IS, Mak MK. Multi-dimensional balance training programme improves balance and gait performance in people with Parkinson's disease: A pragmatic randomized controlled trial with 12-month follow-up. Parkinsonism Relat Disord. 2015 Jun;21(6):615-21. doi: 10.1016/j.parkreldis.2015.03.022. Epub 2015 Mar 31. PMID 25899544
- [Background] Stahl SE, An HS, Dinkel DM, Noble JM, Lee JM. How accurate are the wrist-based heart rate monitors during walking and running activities? Are they accurate enough? BMJ Open Sport Exerc Med. 2016 Apr 25;2(1):e000106. doi: 10.1136/bmjsem-2015-000106. eCollection 2016. PMID 27900173
- [Result] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Result] Steffen T, Seney M. Test-retest reliability and minimal detectable change on balance and ambulation tests, the 36-item short-form health survey, and the unified Parkinson disease rating scale in people with parkinsonism. Phys Ther. 2008 Jun;88(6):733-46. doi: 10.2522/ptj.20070214. Epub 2008 Mar 20. Erratum In: Phys Ther. 2010 Mar;90(3):462. PMID 18356292
- [Result] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Result] Kletzel SL, Hernandez JM, Miskiel EF, Mallinson T, Pape TL. Evaluating the performance of the Montreal Cognitive Assessment in early stage Parkinson's disease. Parkinsonism Relat Disord. 2017 Apr;37:58-64. doi: 10.1016/j.parkreldis.2017.01.012. Epub 2017 Jan 28. PMID 28189463
- [Result] Chaudhuri KR, Martinez-Martin P. Quantitation of non-motor symptoms in Parkinson's disease. Eur J Neurol. 2008 Sep;15 Suppl 2:2-7. doi: 10.1111/j.1468-1331.2008.02212.x. PMID 18702736
- [Result] Li HJ, Zhang MF, Chen MX, Hu AL, Li JB, Zhang B, Liu W. Validation of the nonmotor symptoms questionnaire for Parkinson's disease: results from a Chinese pilot study. Int J Neurosci. 2015;125(12):929-35. doi: 10.3109/00207454.2014.986573. Epub 2014 Dec 18. PMID 25387070
- [Result] Horvath K, Aschermann Z, Acs P, Deli G, Janszky J, Komoly S, Balazs E, Takacs K, Karadi K, Kovacs N. Minimal clinically important difference on the Motor Examination part of MDS-UPDRS. Parkinsonism Relat Disord. 2015 Dec;21(12):1421-6. doi: 10.1016/j.parkreldis.2015.10.006. Epub 2015 Oct 22. PMID 26578041
- [Result] Tsang KL, Chi I, Ho SL, Lou VW, Lee TM, Chu LW. Translation and validation of the standard Chinese version of PDQ-39: a quality-of-life measure for patients with Parkinson's disease. Mov Disord. 2002 Sep;17(5):1036-40. doi: 10.1002/mds.10249. PMID 12360555
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886